CLINICAL TRIAL: NCT01191515
Title: Prospective Evaluation of Near and Intermediate Visual Outcomes With Monofocal Intraocular Lenses: The Mast Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Innovative Medical (Industry)
Collaborators: Staar Surgical Company (Industry)
Responsible Party: Innovative Medical, CRO
Other Study IDs: The Mast Study
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Patients Implanted With Monofocal Intraocular Lens
Keywords: Previous Cataract patients; Monofocal IOL implant; Evaluation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Near visual outcomes with Monofocal IOL: Evaluation of intermediate visual outcomes of patients undergoing routine cataract surgery with phacoemulsification and monofocal IOl placement in the capsular bag in at least one eye.
  Interventions: Device: Monofocal Intraocular Lenses
- Intermediate Visual outcomes: Evaluation of intermediate visual outcomes of patients undergoing routine cataract surgery with phacoemulsification and monofocal IOl placement in the capsular bag in at least one eye.
  Interventions: Device: Monofocal Intraocular Lenses

INTERVENTIONS:
Device: Monofocal Intraocular Lenses — Monofocal Intraocular Lenses

SUMMARY:
The purpose of this study is to evaluate the near and intermediate visual outcomes of patients who have undergone routine cataract surgery (removal of cloudy crystalline lens) with phacoemulsification (the break-up and removal of cloudy lens) and monofocal IOL ( a plastic lens implanted to replace eye's natural lens) placement in the capsular bag in at least one eye.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age
* Patients who underwent routine cataract surgery with phacoemulsification and monofocal iol placement in the capsular bag in at least one eye within the last 36 months
* At least 1 month postop before follow-up evaluation
* All Patients must have a DCVA of 20/25 or better

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective evaluation of 200 patients male or female at least 18 years of age who have previously undergone phacoemulsification (the break-up and removal of a cataract) between one and 36 months earlier
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Campbell, MD, Principal Investigator — Advanced Vision Institute
Locations (1):
- Advanced Vision Institute, Williamsburg, Virginia, United States